CLINICAL TRIAL: NCT00603421
Title: Effectiveness of a 24 Hour Phone Line on the Rate of Suicide Attempts in Borderline Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AOM 05062
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Borderline Personality Disorder
Keywords: borderline personality disorder; suicide; suicidality; suicide attempt; suicidal behavior; self-injurious behavior; self-harm behavior; suicide prevention center; telephone intervention
MeSH Terms: conditions — Borderline Personality Disorder; Suicide; Suicidal Ideation; Suicide, Attempted; Self-Injurious Behavior | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patient benefits from treatment as usual plus access to a crisis 24 hour phone line.
  Interventions: Other: 24 hour phone line
- 2 (Active Comparator): Patient benefits from treatment as usual
  Interventions: Other: treatment as usual

INTERVENTIONS:
Other: 24 hour phone line — 24 hour phone line is available as soon as the patient himself feels necessary. This phone line is supported by professionals of mental health, all specialised in borderline personality disorder
  Arms: 1
Other: treatment as usual — Treatment as usual
  Arms: 2

SUMMARY:
This randomized multicentric clinical trial assesses the effectiveness of 24 hour phone line on the rate of suicide attempts and self-injurious behaviors in borderline patients.

DETAILED DESCRIPTION:
Borderline personality disorder is very frequent among psychiatric populations, and chronic suicidality is a major problem in clinical practice with borderline patients. In a lot of countries, suicide prevention centers are available, but most of these centers are not supervised by professionals of mental health, and none is specifically oriented to the borderline population.

The main goal of this study is to assess the effectiveness of a 24 hour crisis phone line on the rate of suicide attempts in a clinical population of borderline patients (the effectiveness of this phone line access on the rate of self-injurious behaviours will also be studied).

In this multicentric controlled trial, 600 borderline patients (men or women, in or out-patients, between 18 and 40 years-old) are randomized in two arms :

* one with treatment as usual
* one with treatment as usual, PLUS one year of access to a 24 hour crisis phone line (with a team of psychiatrists specialized in borderline personality disorder).

All patients are assessed with standardized instruments (interviewers are blind to the patient's status), at entry (T1) and one year later (T2).

ELIGIBILITY:
Inclusion Criteria:

* 18 to 40 years old
* in or out-patient in one of the recruiting center
* men or women
* with a borderline personality disorder
* written informed consent

Exclusion Criteria:

* inferior to 18 or superior to 40 years old
* schizophrenia
* severe somatic disorder
* participation refusal
* participation to another interventional study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 318 (Actual)
Dates: Start 2009-02; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Rate of suicide attempts | Annual

SECONDARY OUTCOMES:
rate of self injurious behaviors | annual

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Pham-Scottez, MD, Principal Investigator — Centre Hospitalier Sainte Anne
Locations (2):
- France (2):
  - Hôpital St Anne, Paris
  - Hopital Cochin Centre de recherche Clinique Paris Centre, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793